CLINICAL TRIAL: NCT02370160
Title: HM2014-26 DT2219 Immunotoxin for the Treatment of Relapsed or Refractory CD19 (+) and/or CD 22 (+) B-lineage Leukemia or Lymphoma
Brief Title: HM2014-26 DT2219 for Relapsed or Refractory B-Lineage Leukemia or Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014LS093
Record Dates: First submitted 2015-02-18; First posted 2015-02-24 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Refractory B-Lineage Leukemia; Relapsed B-Lineage Leukemia; Refractory B-Lineage Lymphoma; Relapsed B-Lineage Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DT2219ARL (Experimental): A recombinant bispecific antibody-targeted toxin.
  Interventions: Biological: DT2219ARL

INTERVENTIONS:
Biological: DT2219ARL — DT2219ARL at assigned dose IV on day 1, 3, 5, 8 and day 15, 17, 19, and 22. Up to 2 additional courses of DT2219ARL may be given until disease progression and/or unacceptable toxicity.

SUMMARY:
This is a phase I/II study of DT2219 for the treatment of relapsed or refractory CD19 (+) and/or CD 22 (+) B-lineage leukemia and lymphoma. The study consists of two phases - a phase I dose/schedule finding component using the maximum tolerated dose identified during the previous phase I study, but with a higher number of doses and a two-stage phase II extension component to confirm safety and make a preliminary determination of the activity level by disease using the dose identified in phase I.

ELIGIBILITY:
Inclusion Criteria:

* Histologic verification of B-cell lineage leukemia or B cell non-Hodgkin lymphoma and evidence of relapse/refractory disease with the presence of CD19 and/or CD22 by flow cytometry or immunohistochemistry of bone marrow aspirate, peripheral blood or node/tumor biopsy
* Relapsed refractory disease that has failed conventional therapy and other therapies of higher priority
* Karnofsky Performance status of ≥ 60% or, if less than 16 years of age, Lansky Play Score of ≥ 60 (appendix II)
* Recovered from effects of prior therapy
* Peripheral blast count under 50 x 10^9/L
* Adequate organ function within 14 days (30 days for cardiac and pulmonary) of treatment start
* Women of childbearing potential and men should be advised and agree to practice effective methods of contraception during the course of study
* Voluntary written consent with appropriate parent/guardian consent and minor information sheet for participants < 18 years of age

Exclusion Criteria:

* Presence of leukemic or infectious pulmonary parenchymal disease
* Presence of active CNS leukemia
* Presence of any uncontrolled systemic infection
* Documented uncontrolled seizure disorder- a seizure disorder controlled with medication
* Active neurologic disorder - peripheral neuropathy alone does not exclude a patient
* Active Hepatitis B or Hepatitis C (virus detectable by PCR)
* Documented penicillin or cephalosporin allergies
* Pregnant or lactating

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2018-04-08 (Actual); Study Completion 2018-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Bachanova, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DT2219ARL 60 µg/kg/Dose (Phase I); DT2219 80 µg/kg/Dose (Phase I); DT2219 60 µg/kg/Dose (Phase II): A recombinant bispecific antibody-targeted toxin.
  DT2219ARL: DT2219ARL at assigned dose IV on day 1, 3, 5, 8 and day 15, 17, 19, and 22. Up to 2 additional courses of DT2219ARL may be given until disease progression and/or unacceptable toxicity.
Period: Overall Study
Arm/Group | DT2219ARL 60 µg/kg/Dose (Phase I) | DT2219 80 µg/kg/Dose (Phase I) | DT2219 60 µg/kg/Dose (Phase II)
Started | 9 | 6 | 3
Completed | 6 | 2 | 2
Not Completed | 3 | 4 | 1
Not completed — Death | 3 | 4 | 1

BASELINE CHARACTERISTICS:
Arm/Group | DT2219ARL
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.11 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Incidence of Any DLT Attributed to DT2219 in the First Cycle
Description: Dose limiting toxicity (DLT) is defined as any of the following adverse events occurring from study day 1 through 7 days after the last dose of DT2219 of the 1st treatment cycle, and not clearly attributed to the primary malignancy or intercurrent illness:
  * any Grade 5 adverse event
  * any Grade 4 neutropenia or thrombocytopenia lasting more for than 7 days
  * any Grade 3 thrombocytopenia with bleeding
  * any Grade 4 non-hematologic adverse event during DT2219 infusion
  * any Grade 3 non-hematologic adverse event occurring after completion of DT2219 infusion
Time Frame: Day 1 - Day 29
Measure: Number; unit: events
Groups:
- DT2219 (Phase II): A recombinant bispecific antibody-targeted toxin.
  DT2219ARL: DT2219ARL at assigned dose IV on day 1, 3, 5, 8 and day 15, 17, 19, and 22. Up to 2 additional courses of DT2219ARL may be given until disease progression and/or unacceptable toxicity.
Arm/Group | DT2219ARL 60 µg/kg/Dose (Phase I) | DT2219 80 µg/kg/Dose (Phase I) | DT2219 (Phase II)
Number analyzed (Participants) | 9 | 6 | 3
events | 1 | 3 | 0
Statistical Analysis 1: Comparison: DT2219ARL 60 µg/kg/Dose (Phase I) vs DT2219 80 µg/kg/Dose (Phase I); Test type: Other; In Phase I: There were 9 subjects treated on dose level 1 (60 µg/kg/dose). There were 6 subjects treated on Dose level 2 (80 µg/kg/dose). There were four DLT events happened in Phase I. One was treated on dose level 1 and the other three were treated on dose level 2. Therefore the MTD was dose level 1

2. Primary Outcome: Phase ll: Overall Disease Response
Description: Response is defined as complete response, partial response and stable disease. Complete response is defined as the disappearance of all signs of cancer in response to treatment. This does not always mean the cancer has been cured.
  Partial response is defined as a decrease in the size of a tumor, or in the extent of cancer in the body, in response to treatment.
  Stable disease is defined as cancer that is neither decreasing nor increasing in extent or severity.
Time Frame: Day 29
Population: 12 Subjects treated on dose level 1: 4 achieved stable disease and 1 had partial response
Measure: Count of Participants; unit: Participants
Arm/Group | DT2219ARL
Number analyzed (Participants) | 12
Participants | 5

3. Secondary Outcome: Incidence of Serious Adverse Events
Description: A Serious Adverse Event is defined as an adverse event that results in any of the following outcomes:
  * Death
  * A life-threatening adverse event
  * Inpatient hospitalization or prolongation of existing hospitalization
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * A congenital anomaly/birth defect.
  * Important medical event
Time Frame: Day 29
Measure: Number; unit: events
Arm/Group | DT2219ARL 60 µg/kg/Dose (Phase I) | DT2219 80 µg/kg/Dose (Phase I) | DT2219 60 µg/kg/Dose (Phase II)
Number analyzed (Participants) | 9 | 6 | 3
events | 2 | 2 | 1

4. Secondary Outcome: Phase II : Duration of Response
Description: Duration of response was calculated as duration between on-study date and best response date for those patients who achieved complete remission (CR) or partial response (PR)
Time Frame: 1 year
Population: Only 2 participants achieved CR or PR
Measure: Median (Full Range); unit: days
Arm/Group | DT2219ARL
Number analyzed (Participants) | 2
days | 59.5 [27 to 92]

5. Secondary Outcome: Disease-free Survival
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | DT2219ARL 60 µg/kg/Dose (Phase I) | DT2219 80 µg/kg/Dose (Phase I) | DT2219 60 µg/kg/Dose (Phase II)
Number analyzed (Participants) | 9 | 6 | 3
Participants | 7 | 5 | 3

6. Secondary Outcome: Overall Survival
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | DT2219ARL 60 µg/kg/Dose (Phase I) | DT2219 80 µg/kg/Dose (Phase I) | DT2219 60 µg/kg/Dose (Phase II)
Number analyzed (Participants) | 9 | 6 | 3
Participants | 3 | 4 | 2

7. Secondary Outcome: Time to Relapse/Progression
Time Frame: 1 year
Measure: Mean (Full Range); unit: days
Arm/Group | DT2219ARL 60 µg/kg/Dose (Phase I) | DT2219 80 µg/kg/Dose (Phase I) | DT2219 60 µg/kg/Dose (Phase II)
Number analyzed (Participants) | 6 | 3 | 1
days | 27.3 [18 to 36] | 42 [28 to 65] | 30 [30 to 30]

ADVERSE EVENTS:
Time Frame: Day 50 or 30 Days after last dose
Arm/Group | DT2219ARL 60 µg/kg/Dose (Phase I) | DT2219 80 µg/kg/Dose (Phase I) | DT2219 (Phase II)
All-Cause Mortality (participants affected / at risk) | 3/9 | 4/6 | 1/3
Serious Adverse Events (participants affected / at risk) | 2/9 | 2/6 | 1/3
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DT2219ARL 60 µg/kg/Dose (Phase I) (N=9) | DT2219 80 µg/kg/Dose (Phase I) (N=6) | DT2219 (Phase II) (N=3)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DT2219ARL 60 µg/kg/Dose (Phase I) (N=9) | DT2219 80 µg/kg/Dose (Phase I) (N=6) | DT2219 (Phase II) (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 9 (21) | 4 (12) | 3 (3)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (3) | 2 (4)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (5)
Anemia (Blood and lymphatic system disorders) | 6 (12) | 3 (7) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 8 (15) | 5 (13) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 1 (3)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 3 (3) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (3)
Creatinine increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 2 (3) | 1 (1) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (5) | 2 (3) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (3) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 0 (0) | 1 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (10) | 4 (6) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (8) | 3 (4) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4) | 2 (6) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Localized edema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 5 (13) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (4) | 1 (1) | 2 (6)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 6 (8) | 2 (5) | 2 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (3)
Weight gain (Investigations) | 3 (3) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 2 (4) | 2 (4) | 1 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT02370160/Prot_SAP_000.pdf